CLINICAL TRIAL: NCT07404982
Title: Reversal of Spinal Anesthesia Residual Motor Block Via Intrathecal Catheter: A Pilot Study
Brief Title: Reversal of Spinal Anesthesia Residual Motor Block Via Intrathecal Catheter
Acronym: IT-Cath
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Joan Spiegel, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000372
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Joint Replacement Surgery
Keywords: Joint Replacement; Knee Replacement
MeSH Terms: interventions — Saline Solution; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients randomized to the control group will receive a combined spinal intrathecal catheter and the same dosing of spinal medications. All aspects of care and monitoring will be the same as non-study patients. The control group will not receive a dose of intrathecal saline post-op
- Saline administered via the intrathecal catheter (Experimental): Patients randomized to the Intervention group will be administered 10ml of sterile normal saline via the intrathecal catheter post-op prior to catheter removal.
  Interventions: Drug: Normal Saline 10 mL Injection

INTERVENTIONS:
Drug: Normal Saline 10 mL Injection — Patients randomized to this arm will have saline administration via intrathecal catheter post-op prior to removal
  Arms: Saline administered via the intrathecal catheter

SUMMARY:
The purpose of this study is to determine the feasibility of administering a predetermined amount of normal saline into the intrathecal or subarachnoid space via a small spinal catheter to reduce or eliminate the effects of previously injected spinal anesthetic following lower extremity orthopedic surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized, interventional study to assess the feasibility and effectiveness of administering normal saline into the intrathecal or subarachnoid space through a small gauge epidural catheter via a single spinal needle to reverse residual anesthesia following lower extremity orthopedic surgery. This method is adapted from observations in obstetric populations where saline administered via the spinal catheter reduced headaches. This study investigates whether orthopedic patients will also receive unique benefits.

Research procedures overview:

* Randomization to intervention or control arm,
* Use of 6-inch BD 20-gauge Quincke spinal needle, through which a B. Braun Perifix 24-gauge polyurethane catheter
* Administration of normal saline
* Administration of post-operative survey while in the PACU 1 hour
* Follow-up survey 3 days post-surgery
* Medical record review and abstraction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having elective lower extremity joint replacement surgery
2. Patients >18 years

Exclusion Criteria:

1. Contraindications to spinal anesthesia (refusal, lumbar spinal hardware, spinal abnormalities)
2. Patient on anticoagulation not withheld
3. Patient receiving re-operation on the same joint
4. Prior intra-cranial bleeding
5. Patient's ASA status >3
6. Non-English speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time to residual motor blockade reversal | Initiation of spinal anesthetic to reversal, up to sixty minutes after removal of catheter.
  Time to residual motor blockade reversal as measured by Bromage score following saline administration and catheter removal, up to a maximum of 60 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States